CLINICAL TRIAL: NCT03291938
Title: A Phase 1 Study to Evaluate the Safety and Tolerability of IACS-010759 in Subjects With Advanced Solid Tumors and Lymphoma
Brief Title: IACS-010759 in Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0023; NCI-2018-01042 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0023 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Advanced Malignant Solid Neoplasm; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Estrogen Receptor Negative; HER2/Neu Negative; Metastatic Malignant Solid Neoplasm; Pancreatic Ductal Adenocarcinoma; Progesterone Receptor Negative; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8; Recurrent Lymphoma; Refractory Lymphoma; Stage II Pancreatic Cancer AJCC v8; Stage IIA Pancreatic Cancer AJCC v8; Stage IIB Pancreatic Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Triple-Negative Breast Carcinoma; Unresectable Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis; Lymphoma; Pancreatic Neoplasms; Triple Negative Breast Neoplasms | interventions — IACS-010759; Pharmacogenomic Variants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (oxidative phosphorylation inhibitor IACS-010759) (Experimental): INDUCTION PHASE: Patients receive oxidative phosphorylation inhibitor IACS-010759 PO QD on days 1-7 of cycle 1 in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Patients receive oxidative phosphorylation inhibitor IACS-010759 PO QD on days 8 and 15 of cycle 1 and then on days 1, 8, and 15 of subsequent cycles. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Oxidative Phosphorylation Inhibitor IACS-010759; Other: Pharmacodynamic Study; Other: Pharmacokinetic Study

INTERVENTIONS:
Drug: Oxidative Phosphorylation Inhibitor IACS-010759 — Given PO
  Other Names: IACS-010759; OXPHOS Inhibitor IACS-010759
Other: Pharmacodynamic Study — Correlative studies
  Other Names: PHARMACODYNAMIC
Other: Pharmacokinetic Study — Correlative studies
  Other Names: PHARMACOKINETIC; PK Study

SUMMARY:
This phase I trial studies the side effects and best dose of oxidative phosphorylation inhibitor IACS-010759 (IACS-010759) in treating patients with lymphoma that has come back (relapsed) or does not respond to treatment (refractory) or solid tumors that have spread to other places in the body (advanced/metastatic) or cannot be removed by surgery (unresectable). IACS-010759 may stop the growth of cancer or tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of IACS-010759, the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) in subjects with any advanced solid tumor and lymphoma.

SECONDARY OBJECTIVES:

I. To evaluate IACS-010759 pharmacokinetics and preliminary antitumor activity (including overall response rate and duration of response).

EXPLORATORY OBJECTIVES:

I. To evaluate pharmacodynamic and exploratory predictive biomarkers of activity of IACS-010759.

OUTLINE: This is a dose-escalation study.

INDUCTION PHASE: Patients receive oxidative phosphorylation inhibitor IACS-010759 orally (PO) once daily (QD) on days 1-7 of cycle 1 in the absence of disease progression or unacceptable toxicity.

MAINTENANCE PHASE: Patients receive oxidative phosphorylation inhibitor IACS-010759 PO QD on days 8 and 15 of cycle 1 and then on days 1, 8, and 15 of subsequent cycles. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3-6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant.
* Subjects must have histologically confirmed malignancy that is metastatic or unresectable and for which there is no available therapy likely to convey clinical benefit.
* Subjects must have received at least one line of systemic therapy in the advanced/metastatic setting. Subjects with diseases without known effective options are also eligible. a) Subjects with relapsed and/or refractory lymphoma must have had at least 2 prior lines of systemic therapy and are not candidates for high dose therapy/autologous stem cell transplant.
* Subjects must have evaluable disease for the dose escalation, and measurable disease for the dose expansion.
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Subjects must have a life expectancy >= 12 weeks.
* Absolute neutrophil count >= 1,500/mcL.
* Hemoglobin >= 9 g/dL.
* Platelets >= 100,000/mcL.
* Total bilirubin =< 1.5 x the institutional upper limit of normal (ULN).
* Aspartate transaminase (AST) serum glutamic oxaloacetic transaminase (SGOT)/alanine transaminase (ALT) serum glutamic pyruvic transaminase (SGPT) =< 2.5 x institutional ULN or =< 5 x institutional ULN in the presence of liver metastases.
* Creatinine clearance >= 45 mL/min/1.73 m^2 for subjects with creatinine levels above institutional normal.
* Women of childbearing potential (WOCBP) must agree to use an adequate method of contraception during the study and until 3 months after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 3 months after the last treatment. Adequate methods of contraception include: total abstinence when this is in line with the preferred and usual lifestyle of the subject; periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment; male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject.
* Combination of any of the two following (a+b or a+c or b+c): a) use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception; b) placement of an intrauterine device (IUD) or intrauterine system (IUS); c) barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository. In case of use of oral contraception, women should have been stable on the same pill before taking study treatment.
* Oral contraceptives are allowed but should be used in conjunction with a barrier method of contraception due to unknown effect of drug-drug interaction. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
* Subjects must have disease that can be safely biopsied (for RP2D biopsy expansion cohort only), and agree to undergo a pretreatment and on-treatment biopsy.
* Subjects with brain metastases must have completed treatment, either surgery or radiation, 4 weeks or longer prior to screening. A brain magnetic resonance imaging (MRI) demonstrating there is no current evidence of progressive brain metastases is required in subjects with previous brain metastasis. Patients with breast tissue expanders may have brain computerized tomography (CT) for assessment.
* Subjects must not be on full dose oral anticoagulation such as warfarin. Low dose warfarin and prophylactic as well as therapeutic low molecular weight heparin are allowable.
* Subjects who enroll in the triple-negative breast cancer (TNBC) dose expansion cohort should adhere to the American Society for Clinical Pathology (ASCP)/College of American Pathologists (CAP) guidelines for the definition of TNBC.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Subjects who have had chemotherapy or radiotherapy within 3 weeks (4 weeks for immunotherapy; 6 weeks for nitrosoureas or mitomycin C) prior to starting the study agent.
* Subjects with active brain metastases.
* Subjects may not be receiving any other investigational agents or have participated in any other clinical trial involving another investigational agent for treatment of advanced solid tumors or lymphoma within 3 weeks prior to cycle 1, day 1 of the study.
* Subjects who had major surgery or radiation therapy within 4 weeks of the first dose of study drug, except for palliative radiotherapy to a limited field, such as for the treatment of bone pain or a focally painful tumor mass.
* Subjects with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to IACS-010759.
* Subjects receiving metformin or other agents known to increase risk of lactic acidosis.
* Subjects who previously received IACS-010759 or oxidative phosphorylation (OXPHOS) inhibitors.
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active serious bacterial, fungal or viral infection or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects with a history of significant cardiac disease including: congestive heart failure requiring therapy; history of myocardial infarction (MI), angina pectoris, coronary artery bypass graft (CABG) within 6 months prior to starting study treatment; clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade atrioventricular (AV) block (e.g., bifascicular block, Mobitz type II and third degree AV block); left ventricular ejection fraction (LVEF) < 50% evaluated by echocardiogram (ECHO) or multigated acquisition scan (MUGA); increased Fridericia's correction formula (QTcF) (> 450 for men and > 470 for women).
* Women who are breast-feeding or pregnant as evidenced by positive serum or urine pregnancy test performed within 72 hours of first dosing. (Pregnant women are excluded from this study because it is not known whether IACS-010759 has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with IACS-010759 breastfeeding should be discontinued if the mother is treated with IACS-010759.)
* Subjects with significant gastrointestinal abnormalities that may affect absorption (e.g., gastric bypass, short gut syndrome).
* Subjects with known human immunodeficiency virus (HIV), acute chronic hepatitis B virus surface antigen (HBsAg) or hepatitis C virus. (HIV-positive subjects are ineligible because of the potential for pharmacokinetic interactions of antiviral therapy with IACS-010759.)
* Lactic acid levels > 2 mmol/L and/or serum pH < 7.35 at baseline.
* Subjects with other active malignancy in the past 3 years with the exception of adequately treated basal cell or squamous cell carcinoma of the skin, in situ cervical cancer, or another early stage cancer that in the discretion of the investigator(s) is currently in complete remission.
* Subjects with >= Common Terminology Criteria for Adverse Events (CTCAE) grade 2 toxicity (except alopecia) due to prior cancer therapy.
* Subjects with any concomitant disease or condition that, in the clinical judgment of the treating physician, is likely to prevent the subject from complying with any aspect of the protocol or that may put the subject at unacceptable risk.
* Subjects with >= grade 1 peripheral neuropathy at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 2 years
Maximum tolerated dose | Up to day 21

SECONDARY OUTCOMES:
Maximum Plasma concentration of IACS-010759 [Cmax] | Up to 2 years
Overall response rate | Up to 2 years
Duration of response | Up to 2 years

OTHER OUTCOMES:
Pharmacodynamic and predictive biomarkers of activity of IACS-010759 | Up to 2 years
  Blood and tumor samples will be used to assess the pharmacodynamic effects of IACS-010759.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A Yap, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Yap TA, Daver N, Mahendra M, Zhang J, Kamiya-Matsuoka C, Meric-Bernstam F, Kantarjian HM, Ravandi F, Collins ME, Francesco MED, Dumbrava EE, Fu S, Gao S, Gay JP, Gera S, Han J, Hong DS, Jabbour EJ, Ju Z, Karp DD, Lodi A, Molina JR, Baran N, Naing A, Ohanian M, Pant S, Pemmaraju N, Bose P, Piha-Paul SA, Rodon J, Salguero C, Sasaki K, Singh AK, Subbiah V, Tsimberidou AM, Xu QA, Yilmaz M, Zhang Q, Li Y, Bristow CA, Bhattacharjee MB, Tiziani S, Heffernan TP, Vellano CP, Jones P, Heijnen CJ, Kavelaars A, Marszalek JR, Konopleva M. Complex I inhibitor of oxidative phosphorylation in advanced solid tumors and acute myeloid leukemia: phase I trials. Nat Med. 2023 Jan;29(1):115-126. doi: 10.1038/s41591-022-02103-8. Epub 2023 Jan 19. PMID 36658425
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org